CLINICAL TRIAL: NCT06918782
Title: Real-world Experience With Combination Chemotherapy and Osimertinib in Poor Prognostic Group of Metastatic EGFR-mutated Lung Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Chung-Man HO, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Osim-CT1LEGFR
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer (NSCLC)
Keywords: Osimertinib; chemotherapy; ctDNA; advance stage lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination chemotherapy and osimertinib (Experimental): Incorporating chemotherapy with ongoing osimertinib treatment involves initiating osimertinib at the standard dose of 80mg orally once daily. This regimen includes a combination of pemetrexed and carboplatin or cisplatin administered intravenously every 3 weeks for a maximum of 6 cycles, followed by maintenance pemetrexed at a dosage of 500mg/m2 every 3 weeks in cases of non-progressive disease.
  Interventions: Drug: Osimertinib plus platinum doublet chemotherapy

INTERVENTIONS:
Drug: Osimertinib plus platinum doublet chemotherapy — Based on the FLAURA2 study (which was not subdivided into ctDNA clearance subgroups), it is hypothesized that adding systemic chemotherapy to osimertinib will prolong PFS and OS and increase objective response rate even among the poor prognostic subgroup with failed ctDNA clearance after initial osimertinib monotherapy. By incorporating systemic chemotherapy (pemetrexed/carboplatin) to first-line osimertinib treatment among the poor prognostic group of metastatic EGFR-mutant lung adenocarcinoma with failure of plasma ctDNA EGFR mutant clearance despite initial osimertinib treatment.

SUMMARY:
The aims of this study are to determine the potential clinical benefits (in terms of PFS, objective response and OS) of add-on systemic chemotherapy (pemetrexed+carboplatin/cisplatin) to first-line osimertinib treatment among the poor prognostic group of metastatic EGFR-mutant lung adenocarcinoma, i.e. failure of plasma ctDNA EGFR mutant clearance at week 3 after osimertinib treatment

DETAILED DESCRIPTION:
This is a single-arm clinical trial, subjects will be consented prior to the initiation of osimertinib (as per standard-of-care) with baseline plasma ctDNA EGFR mutations tested in QMH. Those with detectable baseline plasma ctDNA EGFR mutations will undergo a repeat plasma ctDNA test after 3 weeks (+/- 5 days) of osimertinib treatment. The screening period is within 42 days. Enrolled eligible subjects will be started on systemic chemotherapy (pemetrexed and carboplatin or cisplatin) within 6 weeks of starting osimertinib, with the following outcome measures:

Primary outcome: real-world 1-year progression-free survival (rw1yPFS) Secondary outcomes: rw response rate (rwRR), rw PFS (rwPFS), rw overall survival (rwOS), rw time-to-treatment discontinuation (rwTTD), ctDNA clearance rate

ELIGIBILITY:
Inclusion Criteria:

1. Adults above 18 years old, both male and female;
2. Pathologically confirmed lung adenocarcinoma with stage IIIB/C or IV disease (TNM staging version 8);
3. Confirmed EGFR common sensitizing mutations (exon 21 L858R or exon 19 del) by locally approved molecular testing methods (allele-specific PCR or NGS) based on tumour tissues or plasma ctDNA;
4. Clinically decided for first-line systemic treatment with osimertinib;
5. Detectable pre-treatment plasma EGFR mutations (by Cobas EGFR Mutation Test v2) and failed clearance 3 weeks (+/- 5 days) after osimertinib treatment;
6. At least one measurable target lesion by RECIST v1.1 criteria;
7. Performance state (ECOG) ≤ 1 and life expectancy ≥ 12 weeks;
8. Females in reproductive age with negative pregnancy test and highly effective means of contraception during and ≥ 4 months after intervention period;
9. Males should agree to have highly effective means of contraception during and ≥ 4 months after intervention period; and
10. Written informed consent obtained.

Exclusion Criteria:

1. Mixed NSCLC and small cell carcinoma;
2. Prior systemic anticancer treatment (targeted therapy, chemotherapy or immunotherapy) for metastatic stage NSCLC;
3. Prior adjuvant chemotherapy or targeted therapy within 6 months;
4. Local radiotherapy within 2 weeks or major surgery within 4 weeks;
5. Inadequate haematological function (haemoglobin < 9 g/dL, neutrophils < 1.5 x 109/L, platelets < 100 x 109/L), renal function (serum creatinine ≥ 1.5 x upper limit of normal (ULN) or creatinine clearance < 45 ml/min) or liver function (total bilirubin > 1.5 x ULN, ALT/AST/ALP > 3 x ULN; ALT/AST/ALP > 5 x ULN for liver metastases; ALP > 5 x ULN for bone metastases);
6. Major medical comorbidities with significant organ dysfunction;
7. Known active hepatitis B or C infection. Chronic hepatitis B on antiviral allowed as per institutional guideline for chemotherapy;
8. Malignancies other than NSCLC; and
9. Known hypersensitivity to pemetrexed or carboplatin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
real-world 1-year progression-free survival | The duration of osimertinib treatment extends from the initiation of therapy until either disease progression or death from any cause, whichever occurs first. Progression-free survival (PFS) will be monitored for up to 1 year.

SECONDARY OUTCOMES:
rw response rate | From date of initiation of osimertinib therapy (day 1) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  real world response rate
OS | From date of initiation of osimertinib therapy (day 1) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  overall survival
rw PFS | The progression-free survival (PFS) will be assessed at the one-year mark.
  real world PFS
rw time-to-treatment discontinuation | From date of initiation of osimertinib therapy (day 1) until the date of first documented discontinuation or date of death from any cause, whichever came first, through study completion, an average of 1 year.
ctDNA clearance rate | The plasma EGFR mutation ctDNA testing will be carried out by Cobas EGFR Mutation Test v2 (Roche Diagnostics) at baseline, 3, 6, 9 and 12 weeks of osimertinib treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James CM Ho, MD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided